CLINICAL TRIAL: NCT01778764
Title: A Comparison of Overall Survival Post-CyberKnife Radiosurgery Treatment of Patients With 1-3 Versus 4 or More Brain Metastases
Brief Title: Phase I Compare OS in Post-CyberKnife Radiosurgery Tx in 1-3 VS 4 or More Brain Metastases
Status: Withdrawn | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Steven D Chang, ROBERT C. AND JEANNETTE POWELL NEUROSCIENCES PROFESSOR, Stanford University
Other Study IDs: IRB-26173; IRB-26173 (Other: Stanford IRB); BRN0022 (Other: OnCore)
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Brain and Nervous System
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- retrospective cohort: retrospective follow-up of patients treated since 2006
- prospective cohort: patients treated over a 5-year period from January 15, 2013 to December 31, 2017 and followed for at least one year thereafter

SUMMARY:
The investigators will learn from this study if the CyberKnife radiosurgery (CK RS) treatment of patients with 1-3 versus 4 or more brain metastases results in the same overall survivals. The importance of this new knowledge will be to determine the treatment efficacy of CK RS with 1-3 versus 4 or more brain metastases. The outcome of this trial would give data to support either the continuation or modification of the CK RS treatment of patients with brain metastases.

DETAILED DESCRIPTION:
This is registry-based cohort study of patients with brain metastases treated at Stanford University Medical Center (SUMC) with CyberKnife radiosurgery (CK RS). It has two components: (1) a retrospective follow-up of patients treated since 2006, and (2) the accrual of a new cohort of patients treated over a 5-year period from January 15, 2013 to December 31, 2017 and followed for at least one year thereafter. The primary aim of this study is to estimate the effect of the number of brain tumor metastases on survival after adjusting for known risk factors for mortality.

ELIGIBILITY:
Inclusion Criteria:

1. the presence of a tumor metastasis or tumor metastases to the brain as manifested by the neurological examination and visibility of the metastatic lesion(s) on MRI and CT scans
2. a Karnofsky performance status (KPS) score of greater than or equal to 60.

Exclusion Criteria:

The exclusion criteria are the converse of the above, i.e. patients without a brain tumor metastasis or brain tumor metastases or a KPS of less than 60.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with all types of primary cancers which have metastasized to the brain.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | until death or the end of follow-up, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chang, Principal Investigator — Stanford University